CLINICAL TRIAL: NCT06577025
Title: A Phase 2, Open-label Study to Evaluate the Efficacy and Safety of Different Sequences of Ciltacabtagene Autoleucel (Cilta-cel), Talquetamab SC in Combination With Daratumumab SC (Tal-D) and Teclistamab SC in Combination With Daratumumab SC (Tec-D) Following Induction With Daratumumab, Bortezomib, Lenalidomide and Dexamethasone (DVRd) in Participants With Standard-risk Newly Diagnosed Multiple Myeloma
Brief Title: A Study of Different Sequences of Cilta-cel, Talquetamab in Combination With Daratumumab and Teclistamab in Combination With Daratumumab Following Induction With Daratumumab, Bortezomib, Lenalidomide and Dexamethasone in Participants With Standard-risk Newly Diagnosed Multiple Myeloma
Acronym: aMMbition
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 54767414MMY2093; 54767414MMY2093 (Other: Janssen Research & Development, LLC); 2023-505792-71-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — talquetamab; daratumumab; Bortezomib; Lenalidomide; Dexamethasone; Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A: DVRd Induction + Tal-D Consolidation + Cilta-cel (Experimental): Participants will undergo apheresis followed by 4 cycles of DVRd induction (each cycle is of 28 days) and cilta-cel will be generated from the participants' T-cells selected from the apheresis product. Upon completion of cilta-cel production, product release, and completion of induction, participants will begin consolidation with 4 cycles of Tal-D (each cycle is of 28 days), followed by a conditioning regimen (cyclophosphamide and fludarabine daily for 3 days); cilta-cel will be administered 5 to 7 days after the start of the conditioning regimen.
  Interventions: Drug: Cilta-cel; Drug: Talquetamab; Drug: Daratumumab; Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone; Drug: Cyclophosphamide; Drug: Fludarabine
- Cohort B: DVRd Induction + Cilta-cel + Tal-D and Tec-D Consolidation (Experimental): Participants will undergo apheresis followed by 4 cycles of DVRd induction and Cilta-cel will be generated from the participants' T-cells selected from the apheresis product. Upon completion of cilta-cel production, product release and completion of induction, participants will begin consolidation with a conditioning regimen (cyclophosphamide and fludarabine daily for 3 days) with infusion of cilta-cel 5 to 7 days after the start of the conditioning regimen. Following cilta-cel infusion, alternating cycles of Tal-D (Cycle 1, 3, 5, and 7) and Tec-D (Cycle 2, 4, 6, and 8) will be started, no earlier than Day 84 and no later than Day 168 post cilta-cel infusion. Each cycle of Tal-D or Tec-D is 84 days which includes an extended treatment-free interval.
  Interventions: Drug: Cilta-cel; Drug: Talquetamab; Drug: Daratumumab; Drug: Teclistamab; Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Drug: Cilta-cel — Cilta-cel infusion will be administered intravenously.
  Other Names: JNJ-68284528, Ciltacabtagene autoleucel
Drug: Talquetamab — Talquetamab will be administered subcutaneously.
  Other Names: JNJ-64407564
Drug: Daratumumab — Daratumumab will be administered subcutaneously as a part of DVRd induction and Tal-D or Tec-D consolidation.
  Other Names: JNJ-54767414
Drug: Teclistamab — Teclistamab will be administered subcutaneously.
  Other Names: JNJ-64007957
  Arms: Cohort B: DVRd Induction + Cilta-cel + Tal-D and Tec-D Consolidation
Drug: Bortezomib — Bortezomib will be administered subcutaneously as a part of induction.
Drug: Lenalidomide — Lenalidomide will be administered orally as a part of induction.
Drug: Dexamethasone — Dexamethasone will be administered orally as a part of induction.
Drug: Cyclophosphamide — Cyclophosphamide will be administered intravenously as a part of conditioning regimen.
Drug: Fludarabine — Fludarabine will be administered intravenously as a part of conditioning regimen.

SUMMARY:
The purpose of this study is to evaluate the rate of response (how effectively treatment is working) with signs of potential cure at 5 years after the start of induction treatment. This is defined as a composite of sustained (at least 2 years) minimal residual disease (MRD) negativity with complete response/stringent complete response (CR/sCR) and a positron emission tomography/computed tomography (PET/CT) scan that does not show any signs of cancer at 5 years. MRD negativity and CR/sCR is defined as no detectable signs of remaining cancer cells after the treatment. This study will also characterize how well the treatments administered work in the study through progression-free survival (PFS). PFS is defined as the length of time during and after the treatment of a disease, that a participant lives with the disease, but it does not get worse.

ELIGIBILITY:
Inclusion Criteria:

* Participants with documented new diagnosis of multiple myeloma (MM) according to international myeloma working group (IMWG) diagnostic criteria and with no prior myeloma-directed therapy
* Participants must have standard-risk MM (stage I and II) based on revised International Staging System (R-ISS)
* Participants must be considered fit (score equals to [=] 0) or intermediate-fit (score=1) according to IMWG Frailty Index assessment (based on the Charlson Comorbidity Index, the Katz Activity of Daily Living and the Lawson Instrumental Activities of Daily Living)
* Measurable disease defined as: Serum monoclonal paraprotein (M-protein) level greater than or equal to (>=) 1.0 gram per deciliter (g/dL) (>=10 gram per liter [g/L] for institutions using alternative units) or urine M-protein level >= 200 milligrams per 24 hours (mg/24 hours); Light chain MM without measurable disease in the serum or the urine: Serum immunoglobulin free light chain >=10 milligrams per deciliter (mg/dL) (>=100 mg/L for institutions using alternative units) and abnormal serum immunoglobulin kappa lambda free light chain ratio
* Eastern Cooperative Oncology Group (ECOG) performance status grade of 0 or 1

Exclusion Criteria:

* Any ongoing myelodysplastic syndrome or B-cell malignancy (other than MM). Any history of malignancy, other than MM, which is considered at high risk of recurrence requiring systemic therapy
* Peripheral neuropathy or neuropathic pain of Grade >= 2, as defined by National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
* Known active or prior history of central nervous system (CNS) involvement or exhibits clinical signs of meningeal involvement of MM
* Stroke or seizure within 6 months of signing the informed consent form (ICF)
* Plasma cell leukemia at the time of diagnosis or any time thereafter through apheresis (>= 5 percent [%] circulating plasma cells in peripheral blood smears), Waldenstrom macroglobulinemia, polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes(POEMS) syndrome, or primary amyloid light chain amyloidosis with associated organ dysfunction
* Presence of high-risk disease features: (a) Cytogenetic high risk lesions by MM fluorescence in situ hybridization (FISH) including deletion 17p (del[17p])/, t(4;14), t(14;16), amplification 1q (amp[1q21]) (>= 4 copies); (b) Presence of 1 or more extramedullary plasmacytomas
* Seropositive for human immunodeficiency virus (HIV)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-09-02 (Estimated)

PRIMARY OUTCOMES:
Rate of Response with Curative Potential | Up to 5 years
  Rate of Response with curative potential is defined as the percentage of participants with a composite of durable (at least 2 years) minimal residual disease (MRD) (10^-5) negativity with complete response/stringent complete response (CR/sCR) by serology and negative positron emission tomography/computed tomography (PET/CT) imaging at 5-years after start of induction therapy. This includes: negative imaging at 5-year landmark time; MRD-negative status (at 10^-5) in 2 bone marrow examinations that are a minimum of 2 years apart; response of CR or better per the International Myeloma Working Group (IMWG) criteria; no examination showing MRD-positive status or relapse from CR in between assessments.
Progression Free Survival (PFS) Rate at 3-Year | At 3-year
  PFS is defined as the time from the date of randomization to either progressive disease (PD), according to the IMWG response criteria, or death, whichever occurs first.
PFS Rate at 5-Year | At 5-year
  PFS is defined as the time from the date of randomization to either PD, according to the IMWG response criteria, or death, whichever occurs first.

SECONDARY OUTCOMES:
Overall response rate (ORR; Partial response [PR] or better) | Up to 5 years
  ORR (PR or better) is defined as the percentage of participants with best overall response of PR or better according to IMWG response criteria.
CR or Better Rate | Up to 5 years
  Rate of CR or better is defined as the percentage of participants with best overall response of CR or better according to IMWG response criteria.
Very Good Partial Response (VGPR) or Better Rate | Up to 5 years
  Rate of VGPR or better is defined as the percentage of participants with best overall response of VGPR or better rate according to IMWG response criteria.
Duration of Response (DOR) | Up to 5 years
  DOR is calculated among responders (with a PR or better response) from the date of initial documented response (PR or better) to the date of first documented evidence of PD as defined according to IMWG criteria or death due to any cause, whichever occurs first.
Time to First Response (TTR) | Up to 5 years
  Time to response (that is, time to first response) is defined as the time between the date of randomization and the first efficacy evaluation that the participant has met all criteria for PR or better based on the computerized algorithm per IMWG criteria for those who had PR or better as their best response.
Duration of CR or Better Response | Up to 5 years
  Duration of CR or better response is calculated among responders (with a CR or better response) from the date of initial documented response CR or better to the date of first documented evidence of PD as defined according to IMWG criteria or death due to any cause, whichever occurs first.
Time to First CR or Better Response | Up to 5 years
  Time to first CR or better response is defined as the time between the date of randomization and the first efficacy evaluation that the participant has met all criteria for CR or better based on the computerized algorithm per IMWG criteria.
PFS on next line therapy (PFS2) | Up to 5 years
  PFS2 is defined as time from randomization to progression on the next line of therapy or death, whichever comes first.
Overall Survival (OS) | Up to 5 years
  OS is measured from the date of randomization to the date of death due to any cause.
MRD-negative CR Rate | Up to 5 years
  MRD-negative CR is defined as the percentage of participants who achieved both CR or better and MRD negativity at a threshold of 10^-5 and 10^-6. MRD-negative CR rate will be evaluated at the first occurrence from induction treatment initiation for participants per IMWG criteria.
Number of Participants with Treatment-emergent Adverse Events (TEAEs) by Severity | Up to 5 years
  An Adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/ biological agent under study. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment. Severity of TEAEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (death). Grade 1= mild, Grade 2= moderate, Grade 3= severe, Grade 4= life-threatening and Grade 5= death related to adverse events.
Change from baseline in Health-related quality of life (HRQoL) (symptoms and functioning) using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Core 30 item instrument (EORTC-QLQ-C30) | Up to 5 years
  Change from baseline in participants' HRQoL (symptoms and functioning) as assessed by EORTC-QLQ-C30 will be reported. The EORTC-QLQ-C30 includes 30 items in 5 functional scales (physical, role, emotional, cognitive, social), 1 global health status scale, 3 symptom scales (pain, fatigue, nausea/vomiting), and 6 single symptom items (dyspnea, insomnia, appetite loss, constipation, diarrhea, financial difficulties). The recall period is 1 week ("past week") and responses are reported using a verbal rating scale. The item and scale scores are transformed to a 0-to-100 scale. A higher score represents greater HRQoL, better functioning, and more (worse) symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (16):
- United States (5):
  - City of Hope, Duarte, California
  - University of California San Francisco, San Francisco, California
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
- Australia (2):
  - Peter MacCallum Cancer Centre, Melbourne
  - The Alfred Hospital, Melbourne
- Brazil (3):
  - Instituto D Or de Pesquisa e Ensino, Salvador
  - Fundacao Antonio Prudente A C Camargo Cancer Center, São Paulo
  - Sociedade Beneficente Israelita Brasileira Hospital Albert Einstein, São Paulo
- Germany (3):
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Tuebingen, Tübingen
  - Universitatsklinikum Wurzburg, Würzburg
- Spain (3):
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Univ. Marques de Valdecilla, Santander

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency